CLINICAL TRIAL: NCT03148561
Title: Misoprostol Versus Expectant Management in Women With Incomplete First-trimester Miscarriage After Misoprostol Treatment: A Randomized Clinical Trial
Brief Title: Management of Women With an Incomplete Miscarriage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MWIE
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Misoprostol group (Other): The women received misoprostol 800 µg (Misotac 200 µg tablets, SIGMA pharmaceutical, Egypt) once dose placed in the posterior vaginal fornix
  Interventions: Drug: Misoprostol
- Expectant group (No Intervention): Women did not receive any medication.

INTERVENTIONS:
Drug: Misoprostol — received misoprostol 800 µg (Misotac 200 µg tablets, SIGMA pharmaceutical) once dose vaginally
  Arms: Misoprostol group

SUMMARY:
Miscarriage is defined as the spontaneous loss of a pregnancy before 24 weeks' gestation, that is, before the fetal viability. The clinical signs of miscarriage are usually vaginal bleeding associated abdominal pain and cramping . The miscarriage is named 'complete' or 'incomplete' according to whether or not tissues are retained in the uterus. If a woman has minimal bleeding but her cervix is closed, this is known as a 'threatened miscarriage. However; if the pregnancy is still inside the uterus but the cervix is open, this is described as an 'inevitable miscarriage', which it will not usually be possible to save the fetus.

From many years, the surgical curettage ('evacuation of the uterus') was considered the 'gold standard management' for miscarriage to remove the retained placental tissue. It is quickly performed and removed almost all the retained products of conception. However, the routine surgical evacuation of the uterus associated with higher rate of morbidity and mortality and should be limited for special indications.

Many studies compared the effectiveness of medical treatment compared to surgery in management of incomplete abortion. There is only one study compared the curettage with expectant management in those women after medical therapy.However; none of them, looked at the effectiveness of the second chance of medical treatment in management of incomplete abortion in trial to avoid the surgical intervention after failure of previous medical treatment. So we think that the immediate evacuation using surgical intervention is truly unnecessary in most cases of failed medical abortion and the patients may get benefit from another trial of medical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Women with confirmed incomplete induced miscarriage, less than 12 weeks' gestation.
2. No known allergy to misoprostol.
3. Women who will be haemodynamically stable.
4. Good access to emergency facilities. Exclusion

1. Women with signs of severe infection ( fever > 38°) 2. Women with severe vaginal bleeding 3. Women known to have allergy to prostaglandins 4. Severe abdominal pain requiring immediate intervention

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
The number of patients with complete miscarriage at 1 week. | 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ali MK, Emam SM, Abdel-Aleem MA, Sobh AMA. Misoprostol versus expectant management in women with incomplete first-trimester miscarriage after failed primary misoprostol treatment: A randomized clinical trial. Int J Gynaecol Obstet. 2021 Sep;154(3):558-564. doi: 10.1002/ijgo.13652. Epub 2021 Mar 24. PMID 33615468